CLINICAL TRIAL: NCT02685475
Title: Comparison of Ultrasound-Guided Axillary Brachial Plexus Block Properties in Diabetic and Non-diabetic Patients: A Prospective Observational Study
Brief Title: Axillary Block Properties in Diabetic Patients
Status: Completed | Type: Observational
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Emine Aysu Salviz, MD, M.D., Attending Anesthesiologist, Istanbul University
Other Study IDs: 2014/1869
Record Dates: First submitted 2016-02-13; First posted 2016-02-18 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2016-03

CONDITIONS: Diabetes Mellitus; Nerve Block Duration; Pain, Postoperative
Keywords: Diabetes mellitus; Axillary brachial plexus block; Block duration; Time-to-first pain; Postoperative analgesia
MeSH Terms: conditions — Diabetes Mellitus; Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Diabetic patients: Patients received ultrasound-guided axillary brachial plexus blocks (ABPBs) with the mixture of 10 mL lidocaine 2% and 20 mL bupivacaine 0.5%.
  Interventions: Drug: Axillary Brachial Plexus Blocks
- Non-diabetic patients: Patients received ultrasound-guided axillary brachial plexus blocks (ABPBs) with the mixture of 10 mL lidocaine 2% and 20 mL bupivacaine 0.5%.
  Interventions: Drug: Axillary Brachial Plexus Blocks

INTERVENTIONS:
Drug: Axillary Brachial Plexus Blocks — All patients received ultrasound-guided axillary brachial plexus block (ABPBs) with the mixture of 10 mL lidocaine 2% and 20 mL bupivacaine 0.5%.
  Other Names: ABPBs

SUMMARY:
Background and objectives: The investigators performed this study to explore whether the presence of diabetes mellitus (DM) would affect the outcomes of axillary brachial plexus blocks (ABPBs) in patients undergoing elective forearm and/or hand surgery. The primary hypothesis was that the sensory block duration would be delayed in diabetic patients.

Methods: After obtaining ethics committee approval and written informed consent, 71 patients were enrolled to the study. Diabetic patients were included in Group DM and non-diabetics were included in Group NODM. All received ultrasound-guided ABPBs with the mixture of 10 mL lidocaine 2% and 20 mL bupivacaine 0.5%. Our primary outcome was sensory block duration, and secondary outcomes were sensory and motor block onset times, motor block duration, time-to-first-pain (numeric rating scale (NRS) ≥4), postoperative NRS scores and rescue analgesic consumption (NRS) ≥4) through the postoperative first 2 days. All outcomes were assessed by a blinded investigators.

DETAILED DESCRIPTION:
Background and objectives: The impact of diabetes mellitus (DM) on the practice of peripheral nerve block anesthesia was mostly investigated in animal researches, and effects on human models are required to be clarified. The investigators performed this study to explore whether the presence of DM would affect the outcomes of axillary brachial plexus blocks (ABPBs) in patients undergoing elective forearm and/or hand surgery. The primary hypothesis was that the sensory block duration would be delayed in diabetic patients.

Methods: After obtaining ethics committee approval and written informed consent, 71 patients with American Society of Anesthesiologists (ASA) physical status I-III and aged between 40 and 75 years were enrolled to the study. Diabetic patients were included in Group DM and non-diabetics were included in Group NODM. All received ultrasound-guided ABPBs with the mixture of 10 mL lidocaine 2% and 20 mL bupivacaine 0.5%. Postoperatively, patients were administered paracetamol as rescue analgesics, if numeric rating scale (NRS) was ≥4. Our primary outcome was sensory block duration, and secondary outcomes were sensory and motor block onset times, motor block duration, time-to-first-pain (numeric rating scale (NRS) ≥4), postoperative NRS scores, and rescue analgesic consumption (NRS) ≥4) through the postoperative first 2 days. All outcomes were assessed by a blinded investigators.

ELIGIBILITY:
Inclusion Criteria:

Patients scheduled for elective forearm and/or hand surgery American Society of Anesthesiologists (ASA) physical status I-III No regional anesthesia contraindication

Exclusion Criteria:

Type 1 DM Type 2 DM patients with only 'diet-controlled' therapy Difficulty with understanding the block and follow-up instructions Significant neurologic disorders Psychiatric or cognitive disorders History of substance abuse Acute and/or chronic opioid use Local anaesthetic hypersensitivity or allergy

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for elective forearm and/or hand surgery
Sampling Method: Non-Probability Sample
Enrollment: 71 (Actual)
Dates: Start 2015-02; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Sensory block duration | 0-24 hours
  Time interval between a successful block and the complete restoration of all the senses controlled by the radial, ulnar, median and musculocutaneous nerves.

SECONDARY OUTCOMES:
Sensory block onset time | 0-30 minutes
  Physical examination with pin-prick test (≥7/8)
Motor block onset time | 0-30 minutes
  Physical examination with modified Bromage scale (≥9/12)
Motor block duration | 0-24 hours
  Time interval between a successful block and the complete restoration of all motor responses controlled by the radial, ulnar, median and musculocutaneous nerves.
Time-to-first pain | 0-48 hours
  Postoperative first pain (NRS ≥4)
Pain (NRS) scores | 0-48 hours
  Numeric rating scale (NRS) pain scores (0: no pain, 10: worst pain imaginable)
Rescue analgesic consumption | 0-48 hours
  Used postoperatively if NRS ≥4

CONTACTS AND LOCATIONS:
Overall Officials: Emine A Salviz, MD, Principal Investigator — Design and conduct the study, review and analyze the data, and write the manuscript
Locations (1):
- Istanbul University, Department of Anesthesiology, Istanbul, Fatih, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gebhard RE, Nielsen KC, Pietrobon R, Missair A, Williams BA. Diabetes mellitus, independent of body mass index, is associated with a "higher success" rate for supraclavicular brachial plexus blocks. Reg Anesth Pain Med. 2009 Sep-Oct;34(5):404-7. doi: 10.1097/AAP.0b013e3181ada58d. PMID 19920415
- [Result] Sertoz N, Deniz MN, Ayanoglu HO. Relationship between glycosylated hemoglobin level and sciatic nerve block performance in diabetic patients. Foot Ankle Int. 2013 Jan;34(1):85-90. doi: 10.1177/1071100712460366. PMID 23386766
- [Result] Cuvillon P, Reubrecht V, Zoric L, Lemoine L, Belin M, Ducombs O, Birenbaum A, Riou B, Langeron O. Comparison of subgluteal sciatic nerve block duration in type 2 diabetic and non-diabetic patients. Br J Anaesth. 2013 May;110(5):823-30. doi: 10.1093/bja/aes496. Epub 2013 Jan 24. PMID 23348203